CLINICAL TRIAL: NCT02664610
Title: REACH OUT: to Reduce High Blood Pressure
Brief Title: Community Study to Reduce High Blood Pressure Through Text Messaging (REACH OUT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lesli E. Skolarus, MD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GO13884
Record Dates: First submitted 2015-10-06; First posted 2016-01-27 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Stroke
Keywords: hypertension treatment; stroke prevention
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No text messages, hypertensive (No Intervention): Participants who have high blood pressure, who are randomized to health information (do not receive text messages).
- Text messages, hypertensive (Experimental): Participants who have high blood pressure, who are randomized to receive text messages.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — hypertensive participants will be randomized to receive tailored, motivational text messages
  Arms: Text messages, hypertensive

SUMMARY:
One of the most powerful predictors of stroke is hypertension, with estimates of approximately 33% of adults in the United States experiencing this condition. Hypertension is significantly more prevalent in African Americans compared to European Americans. Importantly, hypertension is a modifiable stroke risk factor.

This proposal will use a community-based participatory research approach to perform a randomized trial of a mobile phone text-messaging intervention to reduce high blood pressure in an urban African American community in Flint, Michigan.

DETAILED DESCRIPTION:
This is a randomized controlled trial of text messaging and blood pressure self-monitoring to reduce blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 y/o) participants with BP ≥140/90 who have mobile phones with text-messaging capability.

Exclusion Criteria:

* Adult who is illiterate, non-English speaking, pregnant, incarcerated/ institutionalized resident, or has a pre-existing condition that makes follow-up for 6 months unlikely.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesli Skolarus, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Text Messages, Hypertensive | Text Messages, Hypertensive
Started | 46 | 48
Completed | 32 | 41
Not Completed | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Text Messages, Hypertensive | Text Messages, Hypertensive | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.8) | 58 (8.5) | 58 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 47 | 92
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Systolic Blood Pressure
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No Text Messages, Hypertensive | Text Messages, Hypertensive
Number analyzed (Participants) | 32 | 41
mmHg
  Change from baseline | -14.4 (26.4) | -11.3 (22.9)
  Baseline | 162.2 (20.5) | 160.7 (23.6)
  6 months | 146.7 (20.5) | 147.2 (21.8)
Statistical Analysis 1: Comparison: No Text Messages, Hypertensive vs Text Messages, Hypertensive; Test type: Superiority; p = 0.60, t-test, 2 sided

2. Secondary Outcome: Mean Change in Diastolic Blood Pressure
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No Text Messages, Hypertensive | Text Messages, Hypertensive
Number analyzed (Participants) | 32 | 41
mmHg
  Change from baseline | -9.5 (12.9) | -8.6 (15.9)
  Baseline | 99.2 (17.8) | 99.0 (11.8)
  6 months | 88.5 (11.5) | 89.4 (13.9)
Statistical Analysis 1: Comparison: No Text Messages, Hypertensive vs Text Messages, Hypertensive; Test type: Superiority; p = 0.79, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | No Text Messages, Hypertensive | Text Messages, Hypertensive
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48

LIMITATIONS AND CAVEATS:
high lost to follow up rate. Unknown why participants did not complete the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No